CLINICAL TRIAL: NCT07061080
Title: Phase II Study Of Tarlatamab Alone Or In Combination With Chemotherapy In Advanced Neuroendocrine Carcinomas Of The Digestive System Or Unknown Primary Origin
Brief Title: Refractory Advanced diGestive Neuroendocrine Carcinomas Treated With tARlatamab
Acronym: RAGNAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETNE T2419; 2024-514327-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Neuroendocrine Carcinomas of The Digestive System; Advanced Neuroendocrine Carcinomas Unknown Primary Origin
Keywords: Digestive Neuroendocrine carcinomas; Tarlatamab; FOLFIRI; NECs; GEP-NEN

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive: arm A) Tarlatamab or Arm B) Tarlatamab plus FOLFIRI. After the observation of 38 PFS events, an interim analysis will be performed to identify the treatment arm with better PFS and safety outcomes. The decision on which arm should be continued for the second part of the trial will be done taking into account both, PFS and safety profile. The decision will be taken by a scientific committee composed of 4 oncologists. At the time of the interim analysis is expected to have included approximately 54 patients (27 per treatment arm).
  In the second part of the trial, the study will continue recruitment treating all patients with the selected treatment according to the scientific committee . The study will be open until the recruitment of 60 patients in this treatment arm (27 + 33).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Tarlatamab (Active Comparator): Tarlatamab as a standalone treatment through intravenous infusion at 10 mg dose every 14 days (i.e. 2 weeks).
  Interventions: Drug: Tarlatamab
- ARM B: Tarlatamab plus FOLFIRI (Experimental): Tarlatamab as intravenous infusion at 10mg in combination with the standard of care second-line chemotherapy (FOLFIRI)
  Interventions: Drug: Tarlatamab; Drug: standard of care second-line chemotherapy (FOLFIRI)

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab as a standalone treatment through intravenous infusion at 10 mg dose every 14 days (i.e. 2 weeks)
Drug: standard of care second-line chemotherapy (FOLFIRI) — FOLFIRI:: irinotecan intravenously 180 mg/m2 on day 1, followed by 400 mg/m2 folinic acid or 200 mg/m² levofolinate in a 2-h infusion, a 10-min bolus of 400 mg/m2 5-FU, and 2400 mg/m2 5-FU over 46 hours; every 14 days).
  Arms: ARM B: Tarlatamab plus FOLFIRI

SUMMARY:
Neuroendocrine neoplasms (NENs) comprise a heterogeneous family of neoplasms arising from the neuroendocrine cells localized in endocrine glands or from the diffuse neuroendocrine cells such as in the digestive or lung tract.

Treatment for gastroenteropancreatic neuroendocrine tumors (GEP-NEC) is primarily based on chemotherapy regimens, primarily platinum, which achieve limited benefit and a median overall survival of approximately 12 months.

Currently, new treatments that activate the immune system to stimulate antitumor responses and prolong survival in patients with NECs are being investigated.

Given the high levels of DLL3 expression on the cell surface of neuroendocrine tumor cells and its minimal, primarily cytoplasmic, localization in normal tissues, DLL3 is a promising target for the development of T-cell-directed therapies in NECs. Tarlatamab is a HLE BiTE molecule that combines the binding specificities for DLL3 and CD3, which could activate the immune system to fight NEC cells.

The main hypothesis is that treatment with tarlatamab, a bispecific anti-DLL3 and anti-CD3 conjugate, either as a single agent or in combination with standard second-line chemotherapy (FOLFIRI) scheme could be an effective treatment option for patients with advanced neuroendocrine carcinomas of the digestive system or unknown primary origin.

DETAILED DESCRIPTION:
1. RACIONAL Neuroendocrine carcinomas (NECs) are aggressive neoplasms located primarily in the gastroenteropancreatic (GEP) tract or of unknown origin. They are uncommon tumors with an estimated incidence per year that ranges from 5 to 7 cases per 100,000 people. The reported incidence has substantially increased over the last decades, at least partially due to improved diagnostic techniques and clinical awareness.

   Treatment of gastroenteropancreatic neuroendocrine tumors (GEP-NEC) is primarily based on chemotherapy regimens, primarily platinum-based, which achieve limited benefit and a median overall survival of approximately 12 months.

   Dual blockade of PD-1 and CTLA-4 has demonstrated efficacy in several tumor types and achieved prolonged survival in a subset of pretreated patients with Grade 3 GEP-NEN. Therefore, activating the immune system to stimulate antitumor responses and prolong survival in patients with NECs is a feasible strategy to explore. Given the high levels of DLL3 expression on the cell surface of neuroendocrine tumor cells and its minimal, primarily cytoplasmic, localization in normal tissues, DLL3 is a promising target for the development of T-cell-directed therapies in NECs. Tarlatamab is a HLE BiTE molecule that combines the binding specificities for DLL3 and CD3, which could activate the immune system to fight NEC cells. Tarlatamab is currently approved for the treatment of patients with small cell lung cancer.
2. HYPOTHESIS The main hypothesis is that treatment with tarlatamab, a bispecific anti-DLL3 and anti-CD3 conjugate, either as a single agent or in combination with standard second-line chemotherapy (FOLFIRI) scheme could be an effective treatment option for patients with advanced neuroendocrine carcinomas of the digestive system or unknown primary origin.
3. OBJECTIVES

The main objectives:

1. To find the best tarlatamab-based treatment.
2. To evaluate the efficacy of tarlatamab, either as a single agent or in combination with the FOLFIRI regimen, in patients with NECs, assessed in terms of overall survival (OS).

Secondary objectives

1. To evaluate the clinical efficacy results of tarlatamab for patients with NEC.
2. To assess the correlation of risk factors with the efficacy of tarlatamab treatment.
3. To assess the quality of life (QoL) of patients with NEC treated with tarlatamab.
4. To assess the safety of the planned treatment regimen.
5. To determine molecular or clinical predictive biomarkers of response to tarlatamab

4. ENDPOINTS

Primary Endpoint for First Part

The primary endpoint for the first part of this study will be the Progression-free Survival (PFS) rate, defined as the percentage of patients without progression as defined by RECIST V1.1 criteria or death. PFS rate will be calculated for each treatment arm separately once 38 PFS events are reported in the first 54 patients included (27 per treatment arm).

Primary Endpoint for Second Part

The primary endpoint will be the 12-months Overall Survival (OS) rate, defined as the percentage of patients alive after 12 months from the first dose of study treatment. OS will consider death from any cause as an event. Patients alive and free of events at the date of the analysis will be censored at their last known contact. OS will be calculated for each treatment arm separately.

Secondary efficacy endpoints

-Objective response rate (ORR) according to RECIST V1.1 criteria (Appendix 3)

-Disease control rate (DCR).

* Duration of the response (DoR).
* Progression free survival (PFS).
* Overall survival (OS).
* Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3.

Secondary safety endpoints

- Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0

- Frequency of AEs leading to treatment discontinuation.

Secondary translational endpoints

-Blood biomarkers

-Correlation between clinical and molecular determinants and efficacy of tarlatamab

5. STUDY DESIGN

The RAGNAR trial is a two-arm, randomized clinical trial of tarlatamab, either as monotherapy or in combination with standard first-line chemotherapy in patients with NECs. During the first part, patients will be randomized to tarlatamab or tarlatamab plus FOLFIRI. In the second part of the trial, the study will continue enrollment and treat all patients with the regimen chosen in the initial two-arm phase. An initial safety evaluation is planned for the first six patients enrolled in the FOLFIRI + tarlatamab arm to determine if the combination is well tolerated.

Clinic visits will occur on C1D1, C1D8, C1D15, and every 2 weeks ±3 days beginning in cycle 2. Response assessment by computed tomography (CT) or magnetic resonance imaging (MRI) following Response Evaluation Criteria in Solid Tumors (RECIST 1.1) will be performed prior to treatment initiation (baseline), every 8 weeks (+/- 1 week), and every 12 weeks (+/- 2 weeks) thereafter until disease progression, patient withdrawal, initiation of a new line of therapy, or death. Quality of life will be assessed at the baseline and safety visit.

Approximately 87 patients are expected to participate in the study in approximately 10 hospitals in Spain and 10 in France.

6. STUDY POPULATION

Patient with histologically confirmed NEC (Ki-67 >20% or mitotic rate >20 per 10 HPF) of GEP or unknown origin, age ≥18 years, male or female, with unresectable locally advanced or metastatic disease, on second-line treatment after progression to:

i) first-line platinum-based chemotherapy, ii) first-line combination chemotherapy with immunotherapy. Patients must have DLL3-positive tumors, measurable disease per RECIST 1.1, and adequate organ function.

7. TREATMENT

Patients will be randomized 1:1 to receive: arm A) Tarlatamab or Arm B) Tarlatamab plus FOLFIRI. After the observation of 38 PFS events, an interim analysis will be performed to identify the treatment arm with better PFS and safety outcomes. The decision on which arm should be continued for the second part of the trial will be done taking into account both, PFS and safety profile. The decision will be taken by a scientific committee composed of 4 oncologists. At the time of the interim analysis is expected to have included approximately 54 patients (27 per treatment arm).

8. ETHICAL CONSIDERATIONS

The development of new strategies to treat NEC is an unmet need. Patients with NEC have limited therapeutic options, and clinical trials are recommended.

The risks observed with tarlatamab in previous clinical studies are acceptable considering the poor prognosis of patients with NEC and are similar to those described with other treatments. To mitigate these risks, the protocol already includes a gradual intrapatient dose escalation during the first cycle, starting from a low dose of tarlatamab (1 mg). The protocol also considers close monitoring of patients on the day of administration to monitor the potential occurrence of hypersensitivity reactions, CRS, and ICANS. The protocol establishes premedication for the prevention of the most common AEs, including hydration, treatment with dexamethasone or equivalent corticosteroids, and antiemetics for patients treated with FOLFIRI. In addition, the protocol establishes an initial safety cohort composed of the first six patients included in the FOLFIRI + tarlatamab group to determine whether the combination is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent.
2. Patient is ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
4. Histologically confirmed neuroendocrine carcinomas (NECs) of the digestive system or unknown primary origin.

   Note: Carcinomas of pulmonary origin are not eligible.
5. Ki-67 >20% or mitotic rate > 20 per 10 HPF.
6. Metastatic or locally advanced unresectable disease in the second-line treatment, after progression to either:

   1. first-line therapy with platinum-based chemotherapy,
   2. first-line combination of immunotherapy chemotherapy (excluding BITE CD3/DLL3).
7. At least one measurable lesion as defined by RECIST V1.1 (Appendix 3).
8. Only patients with tumors positive for DLL3 as determined by the central laboratory are eligible. DLL3 positivity is defined as ≥1% of DLL3-expressing cells.

   Note: An archival tumor tissue sample (frozen tumor block or 15 unstained formalin fixed, paraffin embedded [FFPE] slides) should be available for submission to the central laboratory for the determination of DLL3. Patients will sign a screening ICF and tumor samples will be sent to the central laboratory for assessing DLL3. Patients who do not have archived tumor tissue available should undergo tumor biopsy.
9. Adequate organ function as defined below

   1. Neutrophil count (ANC) ≥ 1.5 × 109/L.
   2. Platelet count ≥ 100 × 109/L.
   3. Hemoglobin ≥ 9 g/dL.
   4. Prothrombin time (PT)/INR and Partial Thromboplastin Time (PTT) or Activated Partial Thromboplastin Time (APTT) 1.5 x upper limit of normal (ULN). Patients on chronic anticoagulation therapy who do not meet the criteria above may be eligible to enroll after discussion with the medical monitor.
   5. Serum bilirubin ≤ 1.5 × ULN or 2 X ULN for subjects with liver metastases. Note: patients with Gilbert's disease are excluded.
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN or ≤ 5 xULN for patients with liver metastases.
   7. Creatinine clearance (CrCl) ≥ 40 mL/min as estimated by the Cockroft-Gault formula or as measured by 24 hour urine collection (GFR can also be used instead of CrCl) (see Table 10 for Cockcroft-Gault formula).

      10. Female patients must either:

   a. Be of nonchildbearing potential: i. Postmenopausal *(defined as at least 1 year without any menses) prior to screening , or i.i. Documented surgically sterile (e.g.hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion).

   *Those who are amenorrheic due to an alternative medical cause are not considered postmenopausal and must follow the criteria for childbearing potential subjects.

   OR b. If of childbearing potential: i. Agree not to try to become pregnant during the study and for at least 60 days after the last dose of tarlatamab, and 6 months after FOLFIRI.

   i.i.And have a negative urine or serum pregnancy test within 7 days prior to Day 1, i.i.i. And if heterosexually active, agree to abstinence (if in line with the usual preferred lifestyle of the patient) or consistently use a condom plus 1 form of highly effective birth control (Appendix 4) starting at screening and throughout the study period and for 60 days after the last dose of tarlatamab and 6 months after FOLFIRI.

(11) Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for 60 days after the last dose of tarlatamab and 6 months after FOLFIRI.

(12) Male patients must not donate sperm starting at screening and throughout the study period, and for 60 days after the last dose of tarlatamab and 6 months after FOLFIRI.

(13) Male patients with a partner with childbearing potential, or who is pregnant or breastfeeding must agree to abstinence or use a condom plus 1 form of highly effective birth control throughout the study period and for 60 days after the last dose of tarlatamab and 6 months after FOLFIRI.

(14) Patient agrees not to participate in another interventional study while on treatment in the present study.

Exclusion Criteria:

1. The following endocrine tumor types may not be included:

   1. Paraganglioma, adrenal, thyroid parathyroid or pituitary endocrine tumors,
   2. Large or small cell lung neuroendocrine carcinoma of the lung,
   3. Neuroendocrine tumors (NETs) of the gastrointestinal tract or unknown origin (i.e. well differentiated tumors)
2. History of other malignancy within the past 2 years prior to first dose of tarlatamab except:

   1. Malignancy (other than in situ) treated with curative intent and with no known active disease present for 2 years before first dose of tarlatamab and felt to be at low risk for recurrence by the treating physician.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated in situ cancer without evidence of disease.
   4. Prostatic intraepithelial neoplasia without evidence of prostate cancer.
   5. Adequately treated urothelial papillary non-invasive carcinoma.
3. Prior anti-cancer therapy: at least 28 days must have elapsed between any prior anti-cancer therapy and first dose of tarlatamab.
4. Persistence of any toxicity from prior anti-tumor therapy that has not been resolved to grade ≤ 1 (NCI CTCAE V5.0) or to levels dictated in the eligibility criteria.

   Note: exception is made with: i) alopecia; ii) grade ≤ 2 neurotoxicity from platinum based chemotherapy or; iii) irreversible toxicities not otherwise described in the exclusion criteria which are stable for ≥ 21 days after consultation with the medical monitor.
5. Major surgery within 28 days of first dose tarlatamab.
6. Radiation therapy < 2 weeks prior to starting study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
7. Myocardial infarction, and/or symptomatic congestive heart failure (New York Heart Association class II) within 12 months of first dose of tarlatamab.
8. Cardiac ejection fraction < 50%, presence of clinically significant pericardial effusion or clinically significant electrocardiogram findings.
9. History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of first dose of tarlatamab.
10. History of solid organ transplantation.
11. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab.
12. Patients who experienced severe, life-threatening or recurrent (grade 2 or higher) immune-mediated adverse events or infusion-related reactions from previous treatments.
13. Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
14. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
15. History of hypophysitis or pituitary dysfunction.
16. Acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of tarlatamab.
17. Positive tests for Hepatitis B (HBVsAg) or Hepatitis C ribonucleic acid (HCVab) indicating acute or chronic infection.
18. Live and live-attenuated vaccination are prohibited within 28 days prior to the first dose of tarlatamab treatment and for the duration of study.

    Note: Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination should be avoided during screening at least 14 days prior to the first day of tarlatamab treatment. Monkeypox infection vaccination is allowed during the study (except during cycle 1).
19. Patient has known sensitivity and immediate hypersensitivity to any components of tarlatamab or FOLFIRI.
20. Pregnant or breastfeeding patients, and patients planning to become pregnant during the study period and same windows as scheduled for contraceptive measures.
21. History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or medical monitor, if consulted, would pose a risk to subject safety, or interfere with the study evaluation, procedures or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) rate | Throughout the study period, with an average follow-up of 3 years
  The percentage of patients without progression as defined by RECIST V1.1 criteria or death. PFS rate will be calculated for each treatment arm separately once 38 PFS events are reported in the first 54 patients included (27 per treatment arm).
  Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
Overall Survival (OS) rate at 12-months | Throughout the study period, at 12 months from the start of treatment
  Defined as the percentage of patients alive after 12 months from the first dose of study treatment. OS will consider death from any cause as an event. Patients alive and free of events at the date of the analysis will be censored at their last known contact. OS will be calculated for each treatment arm separately. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patient status at each visit according to protocol. Long term follow up to be performed at least every 6 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, with an average follow-up of 3 years
  Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1. This will be considered as the percentage/proportion of patients with complete response (CR) or partial response (PR) as their overall best response throughout the study period. Objective responses will be assessed locally by the investigator according to RECIST, version 1, and indicating the change in size of tumors as compared with baseline, at the first dose of study treatment.
Disease control rate (DCR) | Throughout the study period, with an average follow-up of 3 years
  Assessed locally by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1. DCR will include the percentage/proportion of patients with CR, PR, or SD (maintained > 4 months) as their overall best response throughout the study period. The DCR will be estimated by binomial proportion, dividing the number of patients with CR, PR or SD for at least 4 months for DCR by the total number of patients studied in the population. The corresponding exact 2-sided 95% CIs will be provided. Changes in tumor size from baseline will be calculated and displayed graphically, where appropriate
Duration of response (DoR) | Throughout the study period, with an average follow-up of 3 years
  Time from first response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment. DoR will be summarized using Kaplan-Meier method and displayed graphically, where appropriate. The mean, median DoR and 95% CIs will be provided.
Patient reported health-related quality of life (HRQoL) | Throughout the study period, with an average follow-up of 3 years
  Assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30), version 3. Summary statistics [mean (and SE), median, range and 95% CI] of absolute scores will be reported for all of the subscales of the EORTC QLQ-C30 questionnaire. The mean change of absolute scores from baseline (and 95% CI) will also be assessed. Line charts depicting the means and mean changes of items and subscales over time will be provided.
  The EORTC QLQ-C30 is a questionnaire used to assess the quality of life in cancer patients. It consists of 15 scales, including 5 functional scales, 3 symptom scales, and 9 multi-item and single-item scales for measuring symptoms and global health status. Scores range from 0 to 100, with higher scores indicating better functioning or higher quality of life for functional scales and global health status, but higher scores indicate a higher level of symptoms for symptom scales
Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) | Throughout the study period, with an average follow-up of 3 years
  Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, M.D., Ph.D., Study Chair — Hospital Vall d'hebrón
Locations (19):
- France (8):
  - Brest University Hospital Centre, Brest, Brest
  - Centre Régional de Lutte Contre le Cancer Institut Bergonié (Bordeaux), Bordeaux, Cedex
  - Centre Oscar Lambret, Lille, Lille
  - Hôpital Edouard Herriot (Hospices Civils Lyon), Lyon, Lyon
  - Institut de Cancérologie de l'Ouest (Angers/Nantes), Nantes, Nantes
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Toulouse
  - Institut de Cancérologie de Lorraine (CLCC) Nancy, Vandœuvre-lès-Nancy, Vandœuvre-lès-Nancy Cedex
  - Gustave Roussy, Villejuif, Villejuif,
- Spain (11):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - H.U Germans Trias i Pujols, Badalona, Barcelona
  - H.U. Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario de Burgos (HUBU), Burgos, Burgos
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - H.U Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - H.U La Paz, Madrid, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No